CLINICAL TRIAL: NCT03960944
Title: Psychological Effect of School Based-Yoga on Low-Income School Children: Randomised Controlled Trial
Brief Title: An Experimental Study of Psychological Effect of School Based-Yoga on Low-Income School Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NMP Medical Research Institute (Other)
Collaborators: Arsha Vidya Study Centre (Unknown); United Research International (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: NMP/UNRI
Record Dates: First submitted 2019-05-21; First posted 2019-05-23 (Actual); Last update posted 2019-05-23 (Actual); Status verified 2019-05

CONDITIONS: Psychological Disturbance; Anxiety Disorder of Childhood
MeSH Terms: interventions — Yoga

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Yoga in School Group (Experimental): 30-mins yoga sessions were conducted in schools for 8-weeks
  Interventions: Other: Yoga
- Control Group (No Intervention): Usual Activities in school

INTERVENTIONS:
Other: Yoga — 30 Min Yoga session included of Physical posture, Breathing exercise, Yoga games and Relaxation.
  Arms: Yoga in School Group

SUMMARY:
Poverty is a common experience for many children and families in developing countries. Living in a poor or low-income household has been linked to poor health and increased risk for mental health problems than the general population. Previous studies link psychological well-being with yoga in adolescents and children. This study investigated the effects of a structured yoga program on psychological well-being in low-income school children.

ELIGIBILITY:
Inclusion Criteria:

* Low income Group
* Parental consent to participate in study

Exclusion Criteria:

* Disabilities
* Substance abuse
* Living outside the school areas

Ages: 8 Years to 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 102 (Actual)
Dates: Start 2018-05-21 (Actual); Primary Completion 2018-12-21 (Actual); Study Completion 2019-03-12 (Actual)

PRIMARY OUTCOMES:
Anxiety | Change from baseline to 8 weeks
  Anxiety score was measured through State and Trait Anxiety Inventory

SECONDARY OUTCOMES:
Depression | Changes from baseline to 8 weeks
  Depression Score was measured through Beck Depression Inventory
Self Esteem | Changes from baseline to 8 weeks
  Self Esteem was measured through Rosenberg Self-esteem scale

CONTACTS AND LOCATIONS:
Overall Officials: Buddhatmananda Saraswati, Study Chair — Arsha Vidya Study Centre, India; Divya Gaur, Study Director — United Research International, India; Rajubhai P Odedra, Principal Investigator — NMP Medical Research Institute, India
Locations (3):
- India (3):
  - NMP Medical Research Institute, Mumbai, Maharashtra
  - United Research International, Jaipur, Rajasthan
  - Arsha Vidya Study Centre, Chennai, Tamil Nadu

IPD SHARING:
Plan to Share IPD: Undecided